CLINICAL TRIAL: NCT00495794
Title: Adherence and Intensification of Medications: A Population-Based Clinical Pharmacists Implementation Study Among Hypertensive Diabetes Patients
Brief Title: Adherence and Intensification of Medications (AIM) Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Kaiser Permanente (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDP 06-128; R18DK076622-01 (NIH)
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes; Hypertension
Keywords: diabetes; hypertension; adherence; implementation; medications; organization of care
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist management (Experimental): Eligible patients assigned to - adherence counseling and medication management delivered by a clinical pharmacist trained in behavioral counseling approaches (motivational interviewing)
  Interventions: Behavioral: Clinical pharmacist-based intervention
- Usual care (No Intervention): Eligible patients receive usual care

INTERVENTIONS:
Behavioral: Clinical pharmacist-based intervention — Pharmacist proactive outreach to patients systematically identified as having adherence or intensification problems; their use of tailored adherence counseling strategies; and their authorization to titrate medications according to prespecified algorithms
  Arms: Pharmacist management

SUMMARY:
Background: Good blood pressure (BP) control among patients with diabetes is essential in preventing diabetes complications and has been found to be not only cost-effective but cost-saving. Nonetheless, over 25% of VA patients with diabetes do not have adequate BP control. Among these poorly controlled patients, over 65% have problems with medication adherence or inadequate intensification of medications. We therefore propose a partnership with the VA Pharmacy Benefits Management (PBM) Office and VISN 11 to evaluate a tailored clinical pharmacist-based intervention to improve medication management, adherence and BP control.

Objectives: The specific objectives of this implementation study are: 1) To evaluate the effects of the intervention on blood pressure (primary outcome) and glycemic and lipid control (secondary outcomes); 2) To assess the impact of the intervention on patients' adherence to blood pressure, anti-hyperglycemic, and lipid-lowering regimens, and intensity of these regimens; 3) To evaluate the cost-effectiveness of the intervention compared to usual care; 4) To evaluate the level of attainment of intervention implementation, examine the process of intervention implementation, and determine the potential for sustainability.

DETAILED DESCRIPTION:
Background: Good blood pressure (BP) control among patients with diabetes is essential in preventing diabetes complications and has been found to be not only cost-effective but cost-saving. Nonetheless, over 25% of VA patients with diabetes do not have adequate BP control. Among these poorly controlled patients, over 65% have problems with medication adherence or inadequate intensification of medications. We therefore propose a partnership with the VA Pharmacy Benefits Management (PBM) Office and VISN 11 to evaluate a tailored clinical pharmacist-based intervention to improve medication management, adherence and BP control.

Objectives: The specific objectives of this implementation study are: 1) To evaluate the effects of the intervention on blood pressure (primary outcome) and glycemic and lipid control (secondary outcomes); 2) To assess the impact of the intervention on patients' adherence to blood pressure, anti-hyperglycemic, and lipid-lowering regimens, and intensity of these regimens; 3) To evaluate the cost-effectiveness of the intervention compared to usual care; 4) To evaluate the level of attainment of intervention implementation, examine the process of intervention implementation, and determine the potential for sustainability.

Methods: In this cluster randomized implementation trial, we will proactively identify, using clinical automated data, all diabetes patients within 3 VA sites who have poor blood pressure control and either poor refill adherence or insufficient medication intensification. (NIDDK R18 funds 2 non-VA sites.) Adherence and treatment intensification patterns will also be evaluated for glycemia and lipids if either of these risk factors is poorly controlled. Clinical pharmacists, trained in motivational interviewing techniques and guided by computerized adherence modules, will identify barriers to medication adherence and provide adherence counseling. They will also be authorized to change and titrate medications following site-specific algorithms. Patients in the non-intervention (control) teams will receive usual care. Blood pressure control and refill adherence will be assessed 6-months after the end of the intervention period. We will also conduct a formative evaluation during the course of the study and assess implementation attainment and potential for dissemination.

Status: Data analysis complete. (Enrollment numbers are for VA and non-VA sites [control and intervention].)

ELIGIBILITY:
Inclusion Criteria:

VA inclusion criteria

1. Must be a veteran at a study site;
2. Have a diagnosis of diabetes;
3. Meet blood pressure, medication adherence and intensification requirements (as determined by the study team)

Exclusion Criteria:

VA Exclusion

1. Dementia
2. Traumatic brain injury
3. Pregnancy
4. Age <18 or >100

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4622 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. E. Michele Heisler, MD MPA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Heisler M, Hofer TP, Klamerus ML, Schmittdiel J, Selby J, Hogan MM, Bosworth HB, Tremblay A, Kerr EA. Study protocol: the Adherence and Intensification of Medications (AIM) study--a cluster randomized controlled effectiveness study. Trials. 2010 Oct 12;11:95. doi: 10.1186/1745-6215-11-95. PMID 20939913
- [Result] Klamerus ML, Kerr EA, Bosworth HB, Schmittdiel JA, Heisler M. Characteristics of diabetic patients associated with achieving and maintaining blood pressure targets in the Adherence and Intensification of Medications program. Chronic Illn. 2014 Mar;10(1):60-73. doi: 10.1177/1742395313496590. Epub 2013 Jul 26. PMID 23892775
- [Result] Heisler M, Hofer TP, Schmittdiel JA, Selby JV, Klamerus ML, Bosworth HB, Bermann M, Kerr EA. Improving blood pressure control through a clinical pharmacist outreach program in patients with diabetes mellitus in 2 high-performing health systems: the adherence and intensification of medications cluster randomized, controlled pragmatic trial. Circulation. 2012 Jun 12;125(23):2863-72. doi: 10.1161/CIRCULATIONAHA.111.089169. Epub 2012 May 8. PMID 22570370
- [Result] Meddings J, Kerr EA, Heisler M, Hofer TP. Physician assessments of medication adherence and decisions to intensify medications for patients with uncontrolled blood pressure: still no better than a coin toss. BMC Health Serv Res. 2012 Aug 21;12:270. doi: 10.1186/1472-6963-12-270. PMID 22909303
- [Result] Sussman JB, Zulman DM, Hayward R, Hofer TP, Kerr EA. Cardiac risk is not associated with hypertension treatment intensification. Am J Manag Care. 2012 Aug;18(8):414-20. PMID 22928756
- [Result] Selby JV, Schmittdiel JA, Fireman B, Jaffe M, Ransom LJ, Dyer W, Uratsu CS, Reed ME, Kerr EA, Hsu J. Improving treatment intensification to reduce cardiovascular disease risk: a cluster randomized trial. BMC Health Serv Res. 2012 Jul 2;12:183. doi: 10.1186/1472-6963-12-183. PMID 22747998

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacist Management | Usual Care
Started | 2319 | 2303
Completed | 1797 | 2303
Not Completed | 522 | 0
Not completed — Pharmacist did not activate patient | 522 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist Management | Usual Care | Total
Number analyzed (Participants) | 1797 | 2303 | 4100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.7) | 65.3 (12.1) | 65.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 547 | 721 | 1268
  Male | 1250 | 1582 | 2832
Region of Enrollment [Number; unit: participants]
  United States | 1797 | 2303 | 4100

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Time Frame: 6 months prior to 6 months after the intervention period
Population: intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Pharmacist Management | Usual Care
Number analyzed (Participants) | 1693 | 2162
mmHg | -8.9 [-9.5 to -8.4] | -9.0 [-9.6 to -8.4]

2. Secondary Outcome: A1c Control
Time Frame: 12 months after intervention period
Population: Includes only participants with an A1c in the 12 months after the intervention period.
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Pharmacist Management | Usual Care
Number analyzed (Participants) | 1477 | 1920
percentage of total hemoglobin | 7.4 (1.4) | 7.6 (1.6)

3. Secondary Outcome: LDL Control
Time Frame: 12 months after invention period
Population: Includes only participants with a LDL in the 12 months after the intervention period.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Pharmacist Management | Usual Care
Number analyzed (Participants) | 1410 | 1824
mg/dl | 89.1 (31.1) | 87.8 (32.9)

ADVERSE EVENTS:
Arm/Group | Pharmacist Management | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/2319 | 0/2303
Other Adverse Events (participants affected / at risk) | 0/2319 | 0/2303

LIMITATIONS AND CAVEATS:
In the intervention arm, only 53% of subjects had a pharmacist encounter. Higher rates of participation might have led to a more substantial initial improvement and a detectable longer term effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes